CLINICAL TRIAL: NCT07246343
Title: Impact of Retro-molar Pad Demarcation on Complete Denture Wearers' Satisfaction and Quality of Life: a Cross-over, Double-blind Clinical Trial.
Brief Title: Impact of Retro-molar Pad Demarcation on Complete Denture Wearers' Satisfaction
Acronym: RMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samiha Sartawi (Other)
Collaborators: University of Jordan (Other)
Responsible Party: Sponsor-Investigator, Samiha Sartawi, Principal investigator, University of Jordan
Organization: University of Jordan (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 31/2019-2020; 31/2019-2020 (Other Grant/Funding Number: Deanship of scientific research University of Jordan)
Record Dates: First submitted 2025-09-30; First posted 2025-11-24 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Edentulous Mouth; Quality of Life; Patient Satisfaction; Complete Edentulism; Prosthesis Durability
Keywords: retromolar pad; lower denture; retention; patient satisfaction; quality of life
MeSH Terms: conditions — Mouth, Edentulous; Patient Satisfaction; Prosthesis Failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- edentolous patients (Experimental): patient satisfaction and quality of life
  Interventions: Procedure: carving of retromolar pad area (RMP); Procedure: no carving of the retromolar pad area (RMP)
- Prosthodontist evaluation (Experimental): evaluation of mucosal changes and lower denture retention
  Interventions: Procedure: carving of retromolar pad area (RMP); Procedure: no carving of the retromolar pad area (RMP)

INTERVENTIONS:
Procedure: carving of retromolar pad area (RMP) — carving of the retromolar pad area on the master cat while no carving is done in other studies
Procedure: no carving of the retromolar pad area (RMP) — NO carving of the retromolar pad area (RMP area)

SUMMARY:
the retromolar pad is a critical anatomical landmark in the lower edentulous arch marking the posterior end of any removable prosthesis. The significance of using this area to aid the retention of the lower denture is evaluated in this clinical study especially that the lower denture is always inferior in retention compared to the upper denture as a result of reduced denture bearing area.

DETAILED DESCRIPTION:
The retromolar pad is a key intraoral anatomical landmark in removable prosthodontics. It comprises of non-keratinized loose alveolar tissue covering glandular tissues and muscle fibers. The denture base should extend to cover the retromolar pad. There are variations in the anatomical shape of the retromolar pad, however, no reports in the literature to record that area on the cast and to measure its effect on the retention of the lower denture.

The retromolar pad is a key intraoral anatomical landmark in removable prosthodontics. The denture base should cover the retromolar pad not only to provide proper peripheral seal but also for stability of the denture by adding another plane to resist movements of the base. Furthermore, it remains a stable landmark even in advanced ridge resorption. It is also considered a crucial landmark to determine the occlusal plane where the later terminates posteriorly in the middle of the upper third of the retromolar pad. The mandibular first molar is usually found at the level corresponding to the anterior two thirds of the retromolar pad area. The pad comprises of non-keratinized loose alveolar tissue covering the glandular tissues, fibers of buccinator muscle, fibers of superior constrictor muscle, fibers of ptergomandibular raphe and the terminal part of the tendon of temporalis muscle. After the molars are lost the bone and surrounding soft tissues remodels, resorbs and blends with retromolar pad. The mylohyoid muscles and the buccinator muscles affixed to nearby bony areas are some of the barriers to the chronic but limited bone resorption of the retromalr pad, following tooth loss, time of edentulism, systemic factors, and denture wear.

There are variations in the anatomical shape (pear, triangular and circular) and size of retromolar pad area both in the same patient and in different patients. It was reported that the denture posterior border should be defined at least more posteriorly than in the 2/3 of the retromolar pad (positioned about 7mm distal to the anterior margin of the retromolar pad) and preferably as much as possible to be extended to the distal end dome of the retromolar pad (about 15mm from the anterior margin of the retromolar pad).

The lower denture is usually less retentive than the upper denture due to the reducced surface area covered. The retromolar pad area defines the posterior end of the denture and helps in the retention and stability of the lower denture, however no reports in the literature to record that area on the cast and to measure its effect on retention. Therefore, this clinical study aims to evaluate the effect of carving the retromolar pad area on the retention of the lower denture.

Therefore this clinical study aims to evaluate the effect of carving the retromolar pad area on the retention of lower denture. 50 edentulous patients with no previous denture history will be recruited. Complete dentures will be constructed for each patient with two sets of mandibular dentures by one prosthodontist. One conventional lower denture and one denture with added rertomolar pad whereby one of the dentures will be delivered and after one month the second denture is delivered. Both dentures will be assessed one month after insertion using validated questionnaires. Clinical assessment of the dentures will be performed by two blind prosthodontists on a visual analogue scale. Data will be analyzed using SPSS software.

ELIGIBILITY:
Inclusion Criteria:

* Recent extraction with the last tooth extracted for at least three months ago
* No previous denture experience (first time complete denture wearers) in both maxilla and mandible
* Ridge classification: Atwood's class III in both maxilla and mandible
* No relevant medical conditions or oral pathologies including lesions or ulcers, xerostomia, or tongue tie that could affect the treatment or compliance with treatment
* Both genders aged 40-80 years
* Participants who signed the consent form

Exclusion Criteria:

* denture wearers
* any medical or soft tissue problems
* not signed the consent form

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
patient satisfaction | Two months
  Patient satisfaction after carved and non carved areas in lower denture. After each period, a blinded dentist asked participants to rate their satisfaction on a 100-mm visual analogue scale regarding eating, taste perception, speaking, and phonetics.
patient quality of life | Two months
  The quality of life of participants after carved and non carved areas in lower denture was assessed. Participants were asked to fill the 20-item oral health impact profile for edentulous patients (OHIP-EDENT) before and after treatment with each experimental lower denture.

SECONDARY OUTCOMES:
assessment of mucosal response and denture outcomes. | Two months
  differences in mucosal reaction after using carved denture (CLD) and non carved denture (NCLD) whether presence or absence of redness, erosion, keratosis, ulceration, and denture fissuratum. Two blinded prosthodontists evaluated the CLD and NCLD regarding mucosal changes, and also rated the retention, support, and stability of upper and lower dentures (CLD and NCLD) on a100-mm VAS scale..

CONTACTS AND LOCATIONS:
Overall Officials: SAMIHA SARTAWI, Principal Investigator — University of Jordan
Locations (1):
- University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No
confidentiality of patients

REFERENCES:
- [Background] Sharma A, Deep A, Siwach A, Singh M, Bhargava A, Siwach R. Assessment and Evaluation of Anatomic Variations of Retromolar Pad: A Cross Sectional Study. J Clin Diagn Res. 2016 May;10(5):ZC143-5. doi: 10.7860/JCDR/2016/19551.7880. Epub 2016 May 1. PMID 27437350
- [Background] Bhutta HE, Moharamzadeh K, Martin R, Martin N. Patient Satisfaction with Upper and Lower Complete Dentures: A Service Evaluation Report. Eur J Prosthodont Restor Dent. 2023 Feb 28;31(1):59-71. doi: 10.1922/EJPRD_2416Bhutta13. PMID 35852120

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-08-27): https://cdn.clinicaltrials.gov/large-docs/43/NCT07246343/SAP_000.pdf